CLINICAL TRIAL: NCT06849323
Title: Effect of Su Jok Therapy with Massage and Seed Method on Neck Pain
Brief Title: Effect of Su Jok Therapy on Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/022
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pain; Alternative Medicine; Neck
Keywords: sukok therapy; neck pain; effect
MeSH Terms: conditions — Pain; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): The universe of the study consists of all academic and administrative staff working at a foundation university and suffering from acute neck pain, while the sample will consist of individuals who meet the inclusion criteria. In the power analysis conducted before the study, the Cohen d (0.50) medium value was taken into account for the effect size, and it was calculated that at least 27 people should be included in the study sample to reach at least 80% power at a 95% confidence interval.
  Interventions: Other: Sujok therapy

INTERVENTIONS:
Other: Sujok therapy — The researchers will first detect the pain points in the hands by palpating them with a metal probe, then apply a clockwise massage to the painful point with the same metal probe, and finally complete the intervention by fixing the natural seed. The fixed seed should remain in the area where it is fixed for at least 4-8 hours, it should not come into contact with water or any liquid during this period, and the seed used should be used only once. There should be no wounds/cuts/scratches in the area where the massage and seed are applied, and the tissue integrity should be complete. According to the International Sujok Association (ISA), seeds similar to organs will be used in seed therapy, as well as neutral seeds (fenugreek, buckwheat and mung bean). Buckwheat seed, which is a powerful acupressure, will be applied. The effectiveness of the su jok treatment will be evaluated using the Bournemouth Neck Pain Question on the 11th day after all interventions and as a follow-up after 4 weeks

SUMMARY:
Neck pain, which is a significant problem in modern society, is a multifactorial disease. It negatively affects our lifestyle as well as our lifestyle. It is known that some risk factors such as lack of physical activity, daily computer use, perceived stress and being a woman have an effect on the development of neck pain.

Academicians are among the occupational groups with the highest risk of experiencing chronic neck pain due to factors such as ergonomic conditions and stress.

In a study examining musculoskeletal disorders in academicians, 59% of the participants were found to have complaints of neck pain. In a study conducted by Cagnie et al. with university and office workers, it was reported that the prevalence of neck pain lasting longer than one year was 45.5%, and women were twice as likely to experience neck pain as men. Chronic neck pain is a condition that significantly negatively affects an individual's behavior, quality of life, family and professional life. In addition to all these biopsychosocial effects, neck pain is a serious problem with increased health care costs, decreased work efficiency, and absenteeism. Controlling pain is important for the individual to relax, increase quality of life, and reduce complications. The process can be managed without pharmacological support, which is a cost-effective situation. The aim of pain management is to eliminate pain at the highest level with minimal side effects. There are many different methods that can be used to eliminate or alleviate pain. While pharmacological methods are generally preferred in pain treatment, it is seen that the use of complementary and alternative medicine methods is increasing today. Since nonpharmacological applications in pain treatment are an area where nurses can easily display their independent roles, nurses are also turning to these methods. Su Jok Therapy method, which is the new favorite of an integrated treatment, is also a method used in pain treatment. It was developed by South Korean scientist Professor Park Jae Woo (1942-2010) in 1986. In Korean, "Su" means hand and "Jok" means foot. Su Jok therapy is a modern acupressure/acupuncture that uses the body's independent communication systems on the hands and feet by applying various techniques such as massage, moxa (heating), needle, magnet and seed to the reflection points on the hands and feet. In the literature, it has been revealed that there is a decrease in pain complaints after the application in knee pain, tension-type headache, heel spur, carpal tunnel syndrome syndrome pain. In a study comparing Sujok Therapy and physical therapy in individuals with neck pain, it was found that the pain reduction periods of the patients in the Su Jok group were shorter compared to physical therapy. Cruz et al. reported that 63.3% of those with neck pain had severe pain before the intervention, while 76.6% reported mild pain after the intervention. Studies on the effect of Sujok therapy on neck pain are limited in the literature

DETAILED DESCRIPTION:
The study is a quasi-experimental study and is planned to be conducted in a single group in a pretest-posttest format. Data will be collected face-to-face on a foundation university campus.

The sociodemographic form and the Bournemouth Neck Questionnaire will be used to collect data.

Sociodemographic Form: Participants' age, gender, occupation, smoking, chronic disease status, duration of neck pain, use of non-drug methods to reduce neck pain and drug use will be questioned.

Bournemouth Neck Questionnaire: The Bournemouth Neck Questionnaire is a questionnaire that questions pain intensity, daily social-functional level, anxiety depression level, cognitive and behavioral aspects of fear-avoidance beliefs, and coping with pain. The Bournemouth Neck Questionnaire consists of seven questions and the answers are scored on a numerical analog scale ranging from zero to 10. The maximum score that can be obtained from the questionnaire is 70, and a high score indicates a high level of pain.

Data collection method: Intervention: Each participant will be administered a data collection form and the Bournemouth Neck Questionnaire before the intervention, and then su jok therapy will be applied once a day for 10 days. There will be no additional medical treatment or medication use during the su jok therapy. In practice, although it is stated that the sole of the foot acting as a natural mechanical pressure applicator due to movement increases the effectiveness of the treatment, in field practice, hands are preferred rather than feet due to ease of use. Researchers will first detect pain points in the hands by palpating them with a metal probe, then apply a clockwise massage to the painful point with the same metal probe, and finally complete the intervention by fixing the natural seed. The fixed seed should remain in the area where it is fixed for at least 4-8 hours, it should not come into contact with water or any liquid during this period, and the seed used should be used only once. There should be no wounds/cuts/scratches in the area where the massage and seed are applied, and the tissue integrity should be complete. According to the International Sujok Association (ISA), seeds similar to organs can be used in seed therapy, as well as neutral seeds (fenugreek, buckwheat, and mung bean). In this study, since neck pain will be studied as a musculoskeletal pain, buckwheat seed, which is a powerful acupressure, will be applied. The effectiveness of the su jok treatment will be evaluated using the Bournemouth Neck Pain Questionnaire on the 11th day and 4 weeks later as a follow-up after all interventions.

ELIGIBILITY:
Inclusion Criteria:

Being between 18-64 years of age Having full tissue integrity in the thumbs of both hands and being able to use them actively Being willing to participate in the study Having tension-type and muscle spasm-type neck pain

Exclusion Criteria:

Having undergone any surgical procedure in the cervical region

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Pain change | about four weeks
  A change in the participants' pain is expected to decrease

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jahre H, Grotle M, Smedbraten K, Dunn KM, Oiestad BE. Risk factors for non-specific neck pain in young adults. A systematic review. BMC Musculoskelet Disord. 2020 Jun 9;21(1):366. doi: 10.1186/s12891-020-03379-y. PMID 32517732
- [Background] Cagnie B, Danneels L, Van Tiggelen D, De Loose V, Cambier D. Individual and work related risk factors for neck pain among office workers: a cross sectional study. Eur Spine J. 2007 May;16(5):679-86. doi: 10.1007/s00586-006-0269-7. Epub 2006 Dec 8. PMID 17160393
- [Background] Bolton JE, Humphreys BK. The Bournemouth Questionnaire: a short-form comprehensive outcome measure. II. Psychometric properties in neck pain patients. J Manipulative Physiol Ther. 2002 Mar-Apr;25(3):141-8. doi: 10.1067/mmt.2002.123333. PMID 11986574